CLINICAL TRIAL: NCT04163861
Title: Frequency and Magnitude of Sub-clinical Systolic Dysfunction by Strain Imaging in Heart Failure With Preserved Ejection Fraction
Brief Title: Frequency and Magnitude of Subclinical Systolic Dysfunction by Strain Imaging in Heart Failure With Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Mohamed Mausool Siraj, Principle investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Other Study IDs: 2286
Record Dates: First submitted 2019-03-22; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction
Keywords: Heart failure with preserved ejection fraction; global longitudinal strain; 2D speckle tracking echocardiography; subclinical systolic dysfunction; GLS
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: 31 patients diagnosed as heart failure with preserved ejection fraction per ESC guidelines 2016 on the basis of history, clinical examination and investigations presenting to the department of cardiology, BSMMU were selected inclusion criteria
  1. Patients with regional wall motion abnormality in 2D echocardiography.
  2. Patients with moderate to severe valvular heart diseases.
  3. Patients with prosthetic valves and pacemakers.
  4. Patients with congenital heart diseases.
  5. Patients currently having arrhythmia such as atrial fibrillation on ECG screening during enrollment of patient.
  6. Patients with poor echo window.
  7. Patients who were not interested to take part in the study.
  Interventions: Diagnostic Test: 2d speckle tracking echocardiography; Diagnostic Test: serum BNP level
- 2: 31 normal healthy control subjects of similar age and sex of HFpEF subjects were taken. Normal echocardiograms will be defined as normal LV size and geometry, normal LVEF >55%). patients are free from cardiovascular diseases.
  Interventions: Diagnostic Test: 2d speckle tracking echocardiography

INTERVENTIONS:
Diagnostic Test: 2d speckle tracking echocardiography — 2d speckle tracking echocardiography
Diagnostic Test: serum BNP level — serum BNP level of HFpEF study subjects
  Groups: 1

SUMMARY:
Background: Originally thought to be purely due to LV diastolic dysfunction, studies in western countries have suggested that heart failure with preserved ejection fraction (HFpEF) is more complex. In patients with HFpEF, LV systolic function is commonly considered normal as the global ejection fraction (EF) is normal. However, the EF reflects only the global cardiac contractile function and does not take the subclinical systolic function into consideration. Therefore more attention should be paid on this subset of heart failure population in which the frequency and magnitude of concomitant subclinical systolic dysfunction has not been clearly defined.

Objective: The principal objective of this study was to assess the global longitudinal systolic function of the LV in patients with HFpEF in a tertiary level hospital with the aim of finding out the frequency and magnitude of impaired subclinical systolic dysfunction by using Global Longitudinal Strain (GLS) derived from 2D speckle tracking echocardiography and to see if there is any correlation of GLS with New York Heart Association (NYHA) functional class and BNP level in these patients.

Methods: This was a cross-sectional study conducted from May 2018 to April 2019. A total of 31 patients with HFpEF (Group I) and 31 healthy volunteers of similar age and sex (Group II) were enrolled in the study by consecutive sampling. Detailed history including NYHA functional class, physical examination, relevant investigations including BNP level was done in patients with HFpEF. 2D echocardiography, color Doppler, tissue Doppler and 2D speckle tracking echocardiography was done in both groups. GLS was obtained in a total of 31 patients with HFpEF (Group I), diagnosed according to the 2016 European Society of Cardiology (ESC) guidelines for the diagnosis and treatment of acute and chronic heart failure and compared with GLS of 31 healthy volunteers (Group II), to find out the frequency and magnitude of impaired subclinical systolic function in patients with HFpEF. GLS was also compared with their NYHA functional class and BNP level to find out if any significant relationship is present.

Result: All patients with HFpEF had preserved LV ejection fraction (LVEF>50%) and evidence of diastolic dysfunction. HFpEF patients demonstrated significantly lower GLS compared to healthy controls (14.92 ± 3.16 versus 20.60 ± 1.84). The reduction in LV GLS was statistically significant (p <0.001). Majority of patients with HFpEF (74.2%) had reduced GLS, when reduced GLS was defined as > 2SD below the mean value for healthy volunteers, indicating the presence of subclinical systolic dysfunction in majority of these patients. Worse GLS was associated with higher BNP levels in patients with HFpEF when modeled categorically as quartiles (p = 0.044) and also when modeled continuously (Pearson correlation, r = 0.5, p = 0.004), there was negligible correlation between LV GLS and NYHA symptom class when modeled continuously (Spearman's correlation, rs = 0.052, p = 0.789).

Conclusion: Strain imaging detects impaired systolic function despite preserved global EF in patients with HFpEF. Subclinical systolic dysfunction was frequent in the majority of HFpEF patients. Lower LV GLS is associated with higher BNP level. LV GLS was not associated with NYHA functional class. Further large scale studies are recommended to confirm the findings of this study.

DETAILED DESCRIPTION:
Case: All patients presented with the diagnosis of heart failure with preserved ejection fraction (HFpEF) to Department of Cardiology, BSMMU were initially approached and then selected as case on the basis of inclusion and exclusion criteria. Heart failure diagnosis was made according to the 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. All inclusion criteria were established within 24 hours of presentation. The eligible patients were explained about the study, written informed consent was taken and demographic data were recorded.

Control group: Apparently normal healthy volunteers were initially approached. Medical records were reviewed for prevalent cardiovascular disease (stroke, coronary artery disease, heart failure, arrhythmia), cardiovascular risk factors (hypertension, diabetes mellitus, hyperlipidemia, smoking, renal dysfunction), systemic disease (such as cancer, infections, autoimmune disorders) or any pharmacotherapy Subjects were excluded if any of these were identified. The eligible patients were explained about the study. Written informed consent was taken and demographic data, Pulse, blood pressure and respiratory rate were recorded.

Clinical data, including detailed medical history, cardiovascular risk factors and associated comorbidities of patients with HFpEF were noted. Relevant physical examination was done and recorded in semi-structured designed data collection sheet. Complementary data were collected including chest radiography, ECG, Echocardiography, and relevant laboratory tests. The symptoms of patients were noted. Shortness of breath was graded according to NYHA functional classification. Venous blood samples were collected in plastic vacuum tubes at room temperature for analysis of BNP using chemilumunescent micro particle immunoassay (CMIA) on the ARCHITECT iSystem, on day 1 of presentation in HFpEF cases. Other laboratory investigations including hemoglobin, serum creatinine, HbA1c in diabetics were also done.

Echocardiography was performed by using Vivid E9 (GE Healthcare, Norway) using a 3.5 Mhz transducer. ECG leads were connected before analysis. LV diameters were calculated by M-mode and LVEF by Simpson"s modified biplane method. The LV mass was estimated by using the area length method and adjusted for body surface area. Echocardiographic LV hypertrophy was defined as an LV mass index> 115 g/m2 for men and > 95 g/m2 for women. LV geometry was classified based on relative wall thickness (RWT), defined as (2×diastolic posterior wall thickness)/LV end-diastolic dimension and Left Ventricular Mass Index (LVMi) as recommended by the American Society of Echocardiography (ASE): normal = RWT ≤ 0.42 and no LVH; eccentric hypertrophy = RWT ≤ 0.42 and LVH; concentric remodeling = RWT > 0.42 and no LVH; concentric hypertrophy = RWT > 0.42 and LVH. Right ventricular (RV) function was assessed by tricuspid annular plane systolic excursion (TAPSE) and tricuspid lateral annular systolic velocity (S') by pulsed tissue Doppler. Peak pulmonary arterial systolic pressure (PASP) was estimated as the sum of peak RV-right atrial gradient from the tricuspid valve regurgitant jet and right atrial pressure on the basis of size and collapsibility of inferior vena cava. Presence and severity of valvular heart diseases were assessed by color Doppler imaging and image guided pulsed and continuous Doppler studies according to 2014 AHA/ACC Guidelines for the Management of Patients with Valvular Heart Disease. Patients with more than mild valvular heart diseases were excluded.Diastolic function parameters were measured as follows: peak early diastolic filling (E) and late diastolic filling (A) velocities, E/A ratio, E deceleration time, early diastolic septal and lateral mitral annular velocity (e'), average E/E', peak TR jet velocity, left atrial volume index. Left atrial volume index was calculated using biplane area-length method from apical four and two chamber views at end-systole from the frame preceding mitral valve opening and was indexed to body surface area. Diastolic dysfunction was classified into three grades according to 2016 ASE/EACVI guidelines.

LV longitudinal strains were analyzed by 2D speckle tracking echocardiography for both controls and patients with HFpEF. Cardiac cycles were obtained during a breath hold in end-expiration. Special care was taken to obtain correct view and checking for foreshortening. Endocardial border was traced at end systole, with a frame rate of 50-80/second, from apical long axis, four chambers and two-chambers view. In case of poor tracking, region of interest (ROI) was readjusted. The results of all three planes were combined in a single bull"s eye summary, along with a global longitudinal strain value (GLS) for the LV which was automatically calculated by automated function imaging (AFI). All strain analysis on HFpEF, and normal control subjects was be performed by a single investigator. Two independent investigators analyzed the echocardiography recordings blinded to clinical data. The intra-observer and inter-observer variability of GLS was assessed from 10 randomly selected patients by intra-class correlation coefficient(R). The R value for intra-observer variability was 0.983 and for inter-observer variability was 0.980. This showed good reproducibility of GLS for both same and different operators.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age >18 years) with the diagnosis of heart failure with preserved ejection fraction.
2. Healthy volunteers of similar age and sex distribution as patients with HFpEF.

Exclusion Criteria:

1. Patients with regional wall motion abnormality in 2D echocardiography.
2. Patients with moderate to severe valvular heart diseases.
3. Patients with prosthetic valves and pacemakers.
4. Patients with congenital heart diseases.
5. Patients currently having arrhythmia such as atrial fibrillation on ECG screening during enrollment of patient.
6. Patients with poor echo window.
7. Patients who were not interested to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 31 diagnosed patients with heart failure with preserved ejection fraction 31 normal healthy control subjects with similar age and sex as HFpEF patients
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
frequency and magnitude of subclinical systolic dysfunction in Heartfailure with preserve Title: d ejection fraction patients | 12 months
  Global longitudinal strain value measured in scale by 2d speckle tracking echocardiography correlated with heart failure with preseved ejection fraction patients.LV longitudinal strains were analyzed by 2D speckle tracking echocardiography for both controls and patients with HFpEF. Endocardial border was traced at end systole, with a frame rate of 50-80/second, from apical long axis, four chambers and two-chambers view. The results of all three planes were combined in a single bull"s eye summary, along with a global longitudinal strain value (GLS) for the LV which was automatically calculated by automated function imaging (AFI). All strain analysis on HFpEF, and normal control subjects was be performed by a single investigator. GLS of HFpEF patients and healthy volunteers were compared. reduced GLS in HFpEF was defined as >2SD blow the mean value for healthy volunteers.

SECONDARY OUTCOMES:
relation of GLS with NYHA functional class | 12 months
  relation of GLS with NYHA functional class. NYHA (Ponikowski et al., 2016) New York Heart Association classification of symptoms and physical activity Class I No limitation of physical activity. Ordinary physical activity does not cause undue breathlessness, fatigue, or palpitations.
  Class II Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in undue breathlessness, fatigue, or palpitations.
  Class III Marked limitation of physical activity. Comfortable at rest, but less than ordinary physical activity results in undue breathlessness, fatigue, or palpitations.
  Class IV Unable to carry on any physical activity without discomfort. Symptoms at rest can be present. If any physical activity is undertaken, discomfort is increased.
relation of GLS with BNP level | 12 months
  relation of GLS with BNP level.A serum BNP level >35 pg/ml was considered elevated as per ESC guidelines for management of heart failure 2016.
find out different echocardiographic parameters in heart failure with preserved ejection fraction patients. | 12 months
  find out different echocardiographic parameters in heart failure with preserved ejection fraction patients.
  LV Systolic function, Diastolic function, RV function was assesed.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mausool Siraj, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided